CLINICAL TRIAL: NCT03713398
Title: Improving Mental Health Services for Prisoners With Serious Mental Illnesses
Brief Title: Mental Health Services for Prisoners With SMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-3154; R34MH111855 (NIH)
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Results first posted 2021-09-23 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-08

CONDITIONS: Mental Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T4C-SMI Group (Experimental): Participants will receive the T4C-SMI intervention, in addition to standard prison mental health services
  Interventions: Behavioral: T4C-SMI
- Control Group (No Intervention): The control group receives standard prison mental health services

INTERVENTIONS:
Behavioral: T4C-SMI — T4C-SMI entails a 25-session, manualized intervention that is delivered in a closed-group format at least twice a week over a three-month period. The intervention curriculum includes three modules: nine sessions on social skills training, five sessions on cognitive restructuring activities, and ten sessions on problem-solving methods. Participants assigned to T4C-SMI receive this intervention in addition to any other prison mental health services that they are otherwise eligible to receive during their incarceration.
  Arms: T4C-SMI Group

SUMMARY:
Interventions that address criminogenic risk factors, such as Thinking for a Change (T4C), are not used with prisoners with serious mental illness (SMI) because of the neurocognitive and social impairments associated with SMI. This study examines the effectiveness of T4C with a modified delivery system designed specifically to address the unique needs of persons with SMI in prison, including improving impulsivity, criminal attitudes, and interpersonal problem solving (treatment targets) and levels of aggression, and the amount of behavioral infractions and time spent in administrative segregation in prison (outcomes).

DETAILED DESCRIPTION:
Interventions are urgently needed to improve the delivery and impact of mental health services for persons with serious mental illnesses (SMI) in prison. Treatments addressing the symptoms of mental illness form a critical component of the continuum of services needed by prisoners with SMI. However, a growing body of literature shows that mental health treatments need to be combined with treatments that directly address criminogenic risk factors (i.e., those factors most closely associated with criminal activities). Despite promising evidence, interventions that address criminogenic risk factors, such as Thinking for a Change (T4C), are not used with prisoners with SMI because of the neurocognitive and social impairments associated with SMI. This study examines the effectiveness of T4C with a modified delivery system designed specifically to address the unique needs of persons with SMI in prison. This small-scale randomized controlled trail (RCT) explores the potential effectiveness of T4C-SMI towards improving impulsivity, criminal attitudes, and interpersonal problem solving (treatment targets) and levels of aggression, and the amount of behavioral infractions and time spent in administrative segregation in prison (outcomes). The study will also examine whether the treatment targets for T4C-SMI mediate the intervention's impact on outcomes.

The long-term goal is to grow the evidence-base for interventions with the capacity to improve prison and community-reentry outcomes for persons with SMI. This study will provide the data needed to implement a rigorous RCT in a future study and supports NIMH's mission to develop innovative interventions in mental health services.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* have a diagnosis of schizophrenia, schizoaffective disorder, psychotic disorder, bipolar disorder with psychotic features or major depressive disorder with psychotic features
* have moderate to high risk levels of criminogenic risk factors as determined by the Level of Service and Case Management Inventory (LS/CMI)
* have at least one year or more remaining on their prison sentence at the time of the screening interview

Exclusion Criteria:

* has participated in T4C-SMI within 6 months prior to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Wilson, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- North Carolina Department of Public Safety, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryant FB, Smith BD. Aggression Questionnaire--Short Form. Psyctests. 2001. doi:10.1037/t09754-000
- [Background] D'Zurilla TJ, Nezu AM, Maydeu-Olivares A (n.d). Social Problem-Solving Inventory - Revised. Psyctests. doi:10.1037/t05068-000
- [Background] Mills JF, Kroner DG, Forth AE. Measures of Criminal Attitudes and Associates (MCAA): development, factor structure, reliability, and validity. Assessment. 2002 Sep;9(3):240-53. doi: 10.1177/1073191102009003003. PMID 12216781
- [Background] Patton JH, Stanford MS, Barratt ES. Factor structure of the Barratt impulsiveness scale. J Clin Psychol. 1995 Nov;51(6):768-74. doi: 10.1002/1097-4679(199511)51:63.0.co;2-1. PMID 8778124
- [Background] Stanford MS, Mathias CW, Dougherty DM, Lake SL, Anderson NE, Patton JH. Fifty years of the Barratt Impulsiveness Scale: An update and review. Personality and individual differences. 2009;47(5): 385-395.
- [Background] Raskin A. Discussion: recent developments in ascertainment and scaling of the BPRS. Psychopharmacol Bull. 1988;24(1):122-4. No abstract available. PMID 3387516
- [Background] Shern DL, Wilson NZ, Coen AS, Patrick DC, Foster M, Bartsch DA, Demmler J. Client outcomes II: Longitudinal client data from the Colorado treatment outcome study. Milbank Q. 1994;72(1):123-48. PMID 8164605
- [Derived] Wilson AB, Phillips J, L Villodas M, Parisi A, Dohler E, Ginley C. Assessing the Potential Efficacy of an Intervention for Incarcerated People With Mental Illness. Psychiatr Serv. 2023 Oct 1;74(10):1072-1076. doi: 10.1176/appi.ps.20220355. Epub 2023 Apr 18. PMID 37070261

RESULTS

PARTICIPANT FLOW:
Groups:
- T4C-SMI Group: The research intervention is Thinking for Change for prisoners with mental illness (T4C-MI). This intervention has two components. The first component is Thinking for a Change (T4C), a CBT based group intervention that includes three treatment modules delivered over the course of 25-sessions in a closed-group format to 8-12 people up to twice a week over 12-14 weeks. The second component of T4C-MI is the Targeted Service Delivery Approach (TSDA) that this research team developed for use during the delivery of T4C to compensate for the impact of the neurocognitive and social impairments associated with mental illness on participants' ability to fully engage in and understand T4C's intervention materials.
- Control Group: The control group receives standard prison treatment and programming
Period: Overall Study
Arm/Group | T4C-SMI Group | Control Group
Started | 50 | 50
Completed | 24 | 23
Not Completed | 26 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | T4C-SMI Group | Control Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 0 | 0 | 0
  18 years and older | 50 | 50 | 100
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender was assigned by the prison where the person was incarcerated.
  Participants
    Female | 14 | 14 | 28
    Male | 36 | 36 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 44 | 43 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Cells <5 participants were collapsed into Other/unknown to mitigate deductive disclosure.
  Participants
    Black or African American | 19 | 14 | 33
    White | 16 | 21 | 37
    More than one race | 8 | 9 | 17
    Other/unknown | 7 | 6 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Levels of Aggression Score From Baseline to Month 3
Description: Aggression Questionnaire - Short Form is a 12-item measure with four subscales: physical aggression, verbal aggression, anger, and hostility. Items are scored on a 6-point Likert scale. Scores range from 12 to 72. The higher the score the more aggression present.
Time Frame: Baseline, Month 3
Population: Data not collected for 2 participants
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | T4C-SMI Group | Control Group
Number analyzed (Participants) | 22 | 23
score on a scale | -4.81 (2.34) | -2.68 (2.32)

2. Primary Outcome: Change in Levels of Aggression Score From Baseline to Month 6
Description: as for outcome 1
Time Frame: Baseline, Month 6
Population: Data not collected for 2 participants
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | T4C-SMI Group | Control Group
Number analyzed (Participants) | 22 | 23
score on a scale | -9.16 (2.57) | -5.21 (2.59)

3. Primary Outcome: Number of Participants With Post Test Behavioral Infractions
Description: Number of participants who have at least 1 behavioral infraction following the intervention. Prison records used to ascertain the number of participants who receive behavioral infractions.
Time Frame: End of intervention through Month 9, approximately 6 months total
Measure: Count of Participants; unit: Participants
Arm/Group | T4C-SMI Group | Control Group
Number analyzed (Participants) | 24 | 23
Participants
  Received infraction | 8 | 6
  No infraction | 16 | 17

4. Primary Outcome: Median Number of Days in Administrative Segregation
Description: Prison records will be used to determine the total number of days participants are placed in administrative segregation.
Time Frame: End of intervention through Month 9, approximately 6 months total
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | T4C-SMI Group | Control Group
Number analyzed (Participants) | 24 | 23
Days | 0 [0 to 20] | 0 [0 to 0]

5. Secondary Outcome: Change in Overall Interpersonal Problem Solving Score
Description: The Social Problem Solving Inventory - Revised, Long (SPSI-R:L) is a 52-item measure of problem solving skills and problem orientation. Items are measured on a 5-point Likert scale. It has three subscales: problem orientation, problem solving skills, and social problem-solving inventory. The total raw score range is from 0 to 20. Higher score mean more positive social problem solving skills.
Time Frame: Baseline, Month 3
Population: Data not collected for 3 participants
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | T4C-SMI Group | Control Group
Number analyzed (Participants) | 22 | 22
score on a scale | 1.38 (0.48) | 0.68 (0.48)

6. Secondary Outcome: Change in Overall Criminal Attitudes Score
Description: The Measure of Criminal Attitudes and Associates (MCAA) Part B is a 46-item measure. Responses are recorded in an agree/disagree format. MCAA includes four scales: attitudes toward violence, sentiments of entitlement, antisocial intent, and associates. Scores range from 0 to 46. Lower scores indicate lower levels of criminal attitudes.
Time Frame: Baseline, Month 3
Population: Data not collected for 4 participants
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | T4C-SMI Group | Control Group
Number analyzed (Participants) | 22 | 21
score on a scale | -5.32 (1.56) | -1.68 (1.51)

7. Secondary Outcome: Change in Overall Impulsivity Score
Description: Barratt Impulsiveness Scale (BIS-11) is a 30 item self-report measure. Items scored on a 4-point Likert scale. It is comprised of six subscales including attention, cognitive instability, perseverance, self-control, motor impulsiveness, and cognitive complexity. The total score ranges from 30 to 120. Lower scores indicate lower levels of impulsiveness.
Time Frame: Baseline, Month 3
Population: Data not collected for 3 participants
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | T4C-SMI Group | Control Group
Number analyzed (Participants) | 22 | 22
score on a scale | -7.61 (2.02) | -0.51 (2.03)

ADVERSE EVENTS:
Time Frame: From the signing of the Informed consent up to a total of approximately 9 months afterward.
Arm/Group | T4C-SMI Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT03713398/Prot_SAP_000.pdf